CLINICAL TRIAL: NCT03210155
Title: Effects of Cranial Electrotherapy Stimulation on Psychological Distress and Maternal Functioning in New Mothers During the Postpartum Period
Brief Title: Efficacy of CES in New Mothers During the Post Partum Period
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to change in recruitment site and search team members
Sponsor: Christina Murphey, RN, PhD (Individual)
Responsible Party: Sponsor-Investigator, Christina Murphey, RN, PhD, Associate Professor, Murphey, Christina, RN, PhD
Organization: Murphey, Christina, RN, PhD (Individual)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSRP #36-17
Record Dates: First submitted 2017-06-25; First posted 2017-07-06 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Anxiety; Depression; Insomnia; Sleep Quality
Keywords: Cranial Electrotherapy Stimulation (CES); Efficacy; Post Partum; Anxiety; Depression; Insomnia; Sleep Quality; Maternal Functioning
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The design for the proposed study is a matched-pair, quasi-experimental, 1:1 randomized, double-blind, sham-controlled clinical trial with a longitudinal component. The analytic technique employed to answer the research questions will be repeated measures analysis of covariance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blocked randomization method will be used to assign participants to active and sham groups. Participants will be assigned to CES treatment or sham CES using a 1:1 ratio. Electromedical Products International, Inc. (EPI) will randomize the assignment of appropriate devices to active or sham groups by using a random list of computer generated numbers (1 for active and 2 for sham) in randomly selected block sizes. The PI and participants are blinded to which participants have Alpha-Stim® CES active or sham devices until data analysis is complete. After the completion of data analysis, blinding will be broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Comparator (Active Comparator): About the size of a smart phone, the Alpha-Stim® AID CES device delivers a mild electrical current (100-500 µA) to the brain via ear clips electrodes. The active intervention is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks at 0.5 Hz. 50% duty cycle with a fixed current of 100 µA (subsensory level).
  Interventions: Device: Alpha-Stim AID CES (Active Comparator)
- Sham Comparator (Sham Comparator): The Alpha-Stim® AID CES sham device is identical in appearance to the active device but is inactive and does not emit electrical current to the brain via ear clip electrodes. The sham intervention is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks.
  Interventions: Device: Alpha-Stim AID CES (Sham Comparator)

INTERVENTIONS:
Device: Alpha-Stim AID CES (Active Comparator) — The Alpha-Stim® AID CES device delivers a mild electrical current (100-500 µA) to the brain via ear clips electrodes. The treatment regimen is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks at 0.5 Hz. 50% duty cycle with a fixed current of 100 µA (subsensory level).
  Other Names: Alpha-Stim AID
  Arms: Active Comparator
Device: Alpha-Stim AID CES (Sham Comparator) — The Alpha-Stim® AID CES sham device is inactive and does not emit electrical current to the brain via ear clip electrodes. The sham treatment regimen is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks.
  Other Names: Alpha-Stim AID
  Arms: Sham Comparator

SUMMARY:
The birth of a child is a major life event that can be filled with excitement, anticipation and joy. However, the transition and adaptation to new demands, roles, responsibilities, and changes in relationships can be stressful, especially for new mothers. In addition, new mothers typically encounter physiological changes and struggle with concerns about weight gain, body image, sexuality, and other physical difficulties such as fatigue. These problems may generate or exacerbate stress, lead to an actual or perceived crisis and psychological distress.

Psychological distress, defined as anxiety, depression, and insomnia, in this study, often increases during the postpartum period and can negatively affect maternal mental health status, maternal and family relationships, and infant-child health. The purpose of this study is to evaluate the effects of cranial electrotherapy stimulation (CES) on anxiety, insomnia, depression, and maternal functioning in first time new mothers following childbirth.

DETAILED DESCRIPTION:
The birth of a child is a major life event that can be filled with excitement, anticipation and joy. However, the transition and adaptation to new demands, roles, responsibilities, and changes in relationships can be stressful, especially for first-time mothers. In addition, new mothers typically encounter physiological changes and struggle with concerns about weight gain, body image, sexuality, and other physical difficulties such as fatigue. These problems may generate or exacerbate stress, lead to an actual or perceived crisis and psychological distress.

Psychological distress, defined as depression, anxiety and insomnia, in this study, often increases during the postpartum period and can negatively affect maternal mental health status, maternal and family functioning, and infant-child outcomes. These conditions commonly present as co-morbidities, but are often unrecognized in clinical practice or under-treated as co-morbidities in new mothers. This unrecognized cluster of co-morbidities may lead to psychological distress and subsequently poor outcomes for mothers, their infants and children.

Current treatment recommendations for depression, anxiety and insomnia are primarily pharmaceutical or psychotherapy, both of which have limitations related to cost, time involved and ineffectiveness for some women. Consequently, there is a need to examine other treatment approaches including complementary modalities, such as cranial electrotherapy stimulation (CES), particularly in light of current evidence that shows the efficacy of early detection, intervention and treatment for pregnant and postpartum women.

The primary objective of this study is to investigate the effect of CES on anxiety in new mothers following childbirth. The secondary objectives are to: (1) determine the effects of CES on depression and insomnia; (2) explore the effect of CES on maternal functioning in new mothers following childbirth, and (3) to examine if items 1 & 2 on the 14 item Hamilton Anxiety Rating Scale (HAM-A14) perform well as a screening test for anxiety. Please see the enclosed Instrument Description document for detailed information related to this scale.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a total score of ≥ 16 on the HAM-A14 and ≥2 on both Hamilton Anxiety Rating Scale (HAM-A14) item 1 (anxious mood) and item 2 (tension) at screening and baseline to be considered for inclusion into the study.
2. Participant is a primiparous new mother, 18-45 years inclusive, who had an uncomplicated vaginal or cesarean birth, gave birth to a healthy baby and both mother and baby are healthy at enrollment and randomization in the study.
3. Sexually active female participants of childbearing potential must be self-report practicing, at least, one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female participants of childbearing potential must have a negative urine pregnancy test before receiving study treatment.
4. Written informed consent must be obtained from the participant before study participation.
5. Participant is in good medical health.
6. No current abuse of alcohol or other substance.
7. Capable of giving informed consent.
8. Capable of doing active or sham CES treatments and completing all study requirements independently
9. For compliance, participants need to have completed 85% (36) of treatments to continue participation in the study

Exclusion Criteria:

1. Participant had serious complications during or after a vaginal or cesarean delivery.
2. Participant had multiple births.
3. Participant meets Diagnostic and Statistical Manual of Mental Disorders (DSM)-V criteria for a mental disorder diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by medical history and/or self-report.
4. Participant is clinically judged by the investigator to be at risk for suicide or is acutely suicidal. Participant has attempted suicide one or more times within the past twelve months.
5. Participant has a Hamilton Anxiety Rating Scale (HAM-A14) score above 30 which suggests a very severe clinical level of anxiety symptoms.
6. Participant has a Hamilton Depression Rating Scale (HAM-D17) score above 30 which suggests a very severe clinical level of depressive symptoms.
7. Participant has a psychiatric condition that would require inpatient or partial psychiatric hospitalization.
8. Participant has a significant history of medical disease (i.e. cardiovascular, hepatic (e.g., cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological (seizures), gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
9. Participant is pregnant, planning to become pregnant. If a participant becomes pregnant, she will be dropped from the study immediately and followed appropriately.
10. Participant has had concomitant therapy with another investigational drug, or participation in an investigational drug study within one month before entering this study.
11. Participant has a history of poor compliance or in the investigator's judgment any participant who is not compliant with the requirements of the study.
12. Participant has had previous trial of CES.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Murphey, RN, PhD, Principal Investigator — Texas A&M University - Corpus Christi
Locations (2):
- United States (2):
  - Primay care; OB-GYN Clinic, Austin, Texas
  - Primary care; OB-GYN Clinic, Corpus Christi, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphey C, Carter P, Price LR, Champion JD, Nichols F. Psychological Distress in Healthy Low-Risk First-Time Mothers during the Postpartum Period: An Exploratory Study. Nurs Res Pract. 2017;2017:8415083. doi: 10.1155/2017/8415083. Epub 2017 Jan 16. PMID 28191350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The only subject was recruited from study flyer in May 2018. Subject met inclusion criteria, provided informed consent and was recruited into the study.
Pre-assignment Details: The only subject recruited from study flyer in May 2018. Subject met inclusion criteria, provided informed consent and was recruited into the study.
Period: Overall Study
Arm/Group | Active Comparator | Sham Comparator
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one subject was enrolled and randomly assigned to sham comparator.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Sham Comparator | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1
Number of participants ≥ 10.5 months postpartum [Number; unit: participants] |  | 0 | 0
Delivery criteria [Number; unit: participants] — nominal; yes/no Uncomplicated vag/c-sect birth; Health mother/baby
  participants |  | 1 | 1
Number of subjects who received contraception [Number; unit: participants] — Nominal; yes/no Intrauterine device (IUD); Barrier method in combination with spermicide; oral/hormonal contraception; abstinence
  participants |  | 1 | 1
Number of Participants with No Current Abuse of Alchohol or Other Substance [Number; unit: participants] — Self-report nominal; yes/no Current abuse of alcohol or other substance
  participants |  | 1 | 1
Capable of giving informed consent [Number; unit: participants] — Nominal; yes/no Capable of giving informed consent
  participants |  | 1 | 1
Ability to completing study requirements [Number; unit: participants] — Nominal; yes/no Capable of during active or sham CES treatments and completing all study requirements independently
  participants |  | 1 | 1
Screening instrument criteria [Number; unit: participants] — Initial HAM-A14 items #1 & #2 ≥ 2 Total HAM-A14 score T1 = ≥ 16
  participants |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Rating Scale Scores Over Time
Description: Hamilton Anxiety Rating Scale (HAM-A14):
  The HAM-A probes 14 parameters. Each item is scored on a 5-point scale, ranging from 0=not present to 4=severe and combined to compute a total score. Higher total scores suggest worse outcomes
  Total score: 14-17 = Mild Anxiety Total score: 18-24 = Moderate Anxiety Total score: 25-30 = Severe Anxiety
Time Frame: T1 (Baseline); T2 (3 weeks); T3 (6 Weeks)
Population: No subjects were randomly assigned to an active comparator
Measure: Number; unit: score on a scale
Arm/Group | Active Comparator | Sham Comparator
Number analyzed (Participants) | 0 | 1
score on a scale
  T1 |  | 15
  T2 |  | 15
  T3 |  | 14

2. Secondary Outcome: Hamilton Depression Rating Scale Scores Over Time
Description: Hamilton Depression Rating Scale17 (HAM-D17)
  Although the HAM-D form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe and combined to compute a total score. Nine items are scored from 0-2. Higher total scores suggest worse outcomes.
  Total score: 0-7 = Normal Total score: 8-13 = Mild Depression Total score: 14-18 = Moderate Depression Total score: 19-22 = Severe Depression Total score: ≥ 23 = Very Severe Depression
  8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression Higher total scores suggests worse outcomes
Time Frame: T1 (Baseline); T2 (3 weeks); T3 (6 Weeks)
Population: No subjects were randomly assigned to an active comparator
Measure: Number; unit: score on a scale
Arm/Group | Active Comparator | Sham Comparator
Number analyzed (Participants) | 0 | 1
score on a scale
  T1 |  | 7
  T2 |  | 7
  T3 |  | 8

3. Secondary Outcome: Pittsburgh Sleep Quality Index Scale Scores Over Time
Description: Pittsburg Sleep Quality Index (PSQI19) A 19-item scale that measures sleep quality during the previous month and discriminates between good and poor sleepers The PSQI19 is a 19-item scale that measures sleep quality during the previous month and discriminates between good and poor sleepers 0 = no difficulty 3 = indicates severe difficulty Seven component scores are then added to yield one "global" score, with a range of 0 = 21 points 0 = indicating no difficulty to 21 = indicating severe difficulties in all areas.
Time Frame: T1 (Baseline); T2 (3 weeks); T3 (6 weeks)
Population: No subjects were randomly assigned to an active comparator
Measure: Number; unit: score on a scale
Arm/Group | Active Comparator | Sham Comparator
Number analyzed (Participants) | 0 | 1
score on a scale
  T1 |  | 8
  T2 |  | 7
  T3 |  | 6

4. Secondary Outcome: Insomnia Severity Index Scores Over Time
Description: The Insomnia Severity Index (ISI7) Items include: the severity of sleep onset and maintenance (middle and early morning awakening) difficulties, satisfaction with current sleep pattern, interference with daily functioning, appearance of impairment attributed to the sleep problem, and the degree of concern caused by insomnia
  Total score categories:
  0 - 7 = No clinically significant insomnia 8 - 14 = Sub threshold insomnia 15 - 21 = Clinical insomnia (moderate severity) 22 - 28 = Clinical insomnia (severe) Higher scores indicate worse outcomes
Time Frame: T1 (baseline); T2 (3 weeks); T3 (6 weeks)
Population: No subjects were randomly assigned to an active comparator
Measure: Number; unit: score on a scale
Arm/Group | Active Comparator | Sham Comparator
Number analyzed (Participants) | 0 | 1
score on a scale
  T1 |  | 1
  T2 |  | 2
  T3 |  | 5

5. Secondary Outcome: Barkin Index of Maternal Functioning Scores Over Time
Description: Barkin Index of Maternal Functioning (BIMF20) The Barkin Index of Maternal Functioning (BIMF) is a 20-item self-report measure that was designed to assess overall functioning in the context of new motherhood. After reverse-coding for items 16 and 18, the BIMF is scored by simply summing all 20 items.
  Total score ranges from 0 to 120 Higher scores represent better outcomes
Time Frame: T1 (baseline); T2 (3 weeks); T3 (6 weeks)
Population: No subjects were randomly assigned to an active comparator
Measure: Number; unit: score on a scale
Arm/Group | Active Comparator | Sham Comparator
Number analyzed (Participants) | 0 | 1
score on a scale
  T1 |  | 93
  T2 |  | 97
  T3 |  | 92

ADVERSE EVENTS:
Time Frame: Duration was six weeks.
Description: Definitions do not differ No subjects were randomly assigned to an active comparator
Arm/Group | Active Comparator | Sham Comparator
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Early termination due to change in recruitment site and search team members

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT03210155/Prot_000.pdf